CLINICAL TRIAL: NCT00833014
Title: Dynamic Annuloplasty System With Activation for the Treatment of Mitral Regurgitation
Acronym: DYANA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MiCardia Corporation (Industry)
Responsible Party: Paul Molloy, CEO, MiCardia Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP07-006
Record Dates: First submitted 2009-01-08; First posted 2009-01-30 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental)
  Interventions: Device: Dynamic Annuloplasty Ring (with option to adjust off-pump)

INTERVENTIONS:
Device: Dynamic Annuloplasty Ring (with option to adjust off-pump) — Annuloplasty device repair of mitral valve regurgitation with option to adjust device post implant.

SUMMARY:
The device is a dynamic annuloplasty ring/band that is able to be adjusted in order to correct for mitral regurgitation intraoperatively or postoperatively, off-pump.

ELIGIBILITY:
Inclusion Criteria:

1. This patient requires mitral valve repair with or without concomitant procedures such as coronary artery bypass or another valve reconstruction or replacement.
2. This patient has been diagnosed with a diseased natural valve, based on echocardiography and is a candidate for mitral valve repair.
3. This patient is in satisfactory condition, based on the physical exam and investigator's experience, to be an average or better operative risk. (i.e., likely to survive one year postoperatively).
4. This patient is geographically stable and willing to return to the implant center for follow-up visits.
5. This patient has been adequately informed of his/her participation in the clinical study, and of what will be required of him/her, in order to comply with the protocol.

Exclusion Criteria:

1. This patient is less than eighteen (18) years of age.
2. This patient has a non-cardiac major or progressive disease, which in the investigator's experience produces an unacceptable increased risk to the patient, or results in a life expectancy of less than twelve months.
3. This patient has an ejection fraction < 30%.
4. This patient has a heavily calcified annulus or leaflets.
5. This patient presents with active endocarditis or has had active endocarditis in the last 3 months.
6. This patient is pregnant (urine HCG test result positive) or lactating.
7. This patient is an intravenous drug abuser or alcohol abuser.
8. This patient has a previously implanted prosthetic mitral valve.
9. This patient requires mitral valve replacement.
10. This patient has a creatinine level > 2.0 mg/dl
11. This patient has had congestive heart failure within the past 6 months requiring surgical treatment.
12. This patient has had a coronary artery ischemic event within the past 6 months.
13. This patient has a known life threatening, non-cardiac disease that will limit the patient's life expectancy to less than one year.
14. This patient is unable to take Coumadin.
15. This patient has a known untreatable allergy to contrast media or nickel.
16. This patient has had a cerebral vascular event within the past 6 months.
17. This patient is a prisoner (U.S.A. Only).
18. This patient is participating in concomitant research studies of investigational products.
19. This patient will not agree to return to the implant center for the required number of follow-up visits or is geographically unavailable for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from major complications and SAM (Systolic Anterior Motion) | 6 months

SECONDARY OUTCOMES:
Ability to adjust annuloplasty ring off-pump post implantation to correct for residual regurgitation, reduction of mitral valve regurgitation at follow-up visits (discharge, 30 days, 6 months) | 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- University of British Columbia, Vancouver, British Columbia, Canada
- Germany (3):
  - University of Saarlands, Homburg
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - University of Leipzig Herzzentrum, Leipzig
- Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- [Background] Baev B, Petkov D, Iliev R, Nachev G. [Mitral valve repair for mitral regurgitation--15 year results]. Khirurgiia (Sofiia). 2006;(4-5):19-22. Bulgarian. PMID 18843917
- [Background] Manesis EK, Cameron CH, Gregoriadis G. Hepatitis-B-surface-antigen-containing liposomes enhance humoral and cell-mediated immunity to the antigen [proceedings]. Biochem Soc Trans. 1979 Aug;7(4):678-80. doi: 10.1042/bst0070678. No abstract available. PMID 225223
- [Background] McGee EC, Gillinov AM, Blackstone EH, Rajeswaran J, Cohen G, Najam F, Shiota T, Sabik JF, Lytle BW, McCarthy PM, Cosgrove DM. Recurrent mitral regurgitation after annuloplasty for functional ischemic mitral regurgitation. J Thorac Cardiovasc Surg. 2004 Dec;128(6):916-24. doi: 10.1016/j.jtcvs.2004.07.037. PMID 15573077
- [Background] Sharony R, Saunders PC, Nayar A, McAleer E, Galloway AC, Delianides J, Schwartz CF, Applebaum RM, Kronzon I, Colvin SB, Grossi EA. Semirigid partial annuloplasty band allows dynamic mitral annular motion and minimizes valvular gradients: an echocardiographic study. Ann Thorac Surg. 2004 Feb;77(2):518-22; discussion 522. doi: 10.1016/j.athoracsur.2003.06.005. PMID 14759429
- [Background] Hashim SW, Rousou AJ, Geirsson A, Ragnarsson S. Solving the puzzle of chronic ischemic mitral regurgitation. Yale J Biol Med. 2008 Dec;81(4):167-73. PMID 19099047
- [Background] Leacche M, Balaguer JM, Byrne JG. Role of cardiac surgery in the post-myocardial infarction patient with heart failure. Curr Heart Fail Rep. 2008 Dec;5(4):204-10. doi: 10.1007/s11897-008-0031-z. PMID 19032915
- [Background] Spoor MT, Bolling SF. Valve pathology in heart failure: which valves can be fixed? Heart Fail Clin. 2007 Jul;3(3):289-98. doi: 10.1016/j.hfc.2007.04.008. PMID 17723937
- [Background] Bolling SF. Mitral reconstruction in cardiomyopathy. J Heart Valve Dis. 2002 Jan;11 Suppl 1:S26-31. PMID 11843517
- [Background] Lloyd-Jones D, Adams R, Carnethon M, De Simone G, Ferguson TB, Flegal K, Ford E, Furie K, Go A, Greenlund K, Haase N, Hailpern S, Ho M, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott M, Meigs J, Mozaffarian D, Nichol G, O'Donnell C, Roger V, Rosamond W, Sacco R, Sorlie P, Stafford R, Steinberger J, Thom T, Wasserthiel-Smoller S, Wong N, Wylie-Rosett J, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2009 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2009 Jan 27;119(3):e21-181. doi: 10.1161/CIRCULATIONAHA.108.191261. Epub 2008 Dec 15. No abstract available. PMID 19075105
- [Background] Liddicoat JR, Mac Neill BD, Gillinov AM, Cohn WE, Chin CH, Prado AD, Pandian NG, Oesterle SN. Percutaneous mitral valve repair: a feasibility study in an ovine model of acute ischemic mitral regurgitation. Catheter Cardiovasc Interv. 2003 Nov;60(3):410-6. doi: 10.1002/ccd.10662. PMID 14571496
- [Background] Bursi F, Enriquez-Sarano M, Nkomo VT, Jacobsen SJ, Weston SA, Meverden RA, Roger VL. Heart failure and death after myocardial infarction in the community: the emerging role of mitral regurgitation. Circulation. 2005 Jan 25;111(3):295-301. doi: 10.1161/01.CIR.0000151097.30779.04. Epub 2005 Jan 17. PMID 15655133
- [Background] Badhwar V, Bolling SF. Mitral valve surgery in the patient with left ventricular dysfunction. Semin Thorac Cardiovasc Surg. 2002 Apr;14(2):133-6. doi: 10.1053/stcs.2002.32314. PMID 11988951
- [Background] Pfeffer MA, Braunwald E. Ventricular remodeling after myocardial infarction. Experimental observations and clinical implications. Circulation. 1990 Apr;81(4):1161-72. doi: 10.1161/01.cir.81.4.1161. PMID 2138525
- [Background] Gillinov AM, Cosgrove DM 3rd. Current status of mitral valve repair. Am Heart Hosp J. 2003 Winter;1(1):47-54. doi: 10.1111/j.1541-9215.2003.02082.x. PMID 15785176
- [Background] Moss RR, Humphries KH, Gao M, Thompson CR, Abel JG, Fradet G, Munt BI. Outcome of mitral valve repair or replacement: a comparison by propensity score analysis. Circulation. 2003 Sep 9;108 Suppl 1:II90-7. doi: 10.1161/01.cir.0000089182.44963.bb. PMID 12970215
- [Background] Ling LH, Enriquez-Sarano M, Seward JB, Tajik AJ, Schaff HV, Bailey KR, Frye RL. Clinical outcome of mitral regurgitation due to flail leaflet. N Engl J Med. 1996 Nov 7;335(19):1417-23. doi: 10.1056/NEJM199611073351902. PMID 8875918
- [Background] Tanemoto K. Surgical treatment of ischemic mitral valve regurgitation. Ann Thorac Cardiovasc Surg. 2005 Aug;11(4):228-31. PMID 16148868
- [Background] Le HC, Thys DM. Ischemic mitral regurgitation. Semin Cardiothorac Vasc Anesth. 2006 Mar;10(1):73-7. doi: 10.1177/108925320601000113. PMID 16703238
- [Background] Gillinov AM, Cosgrove DM 3rd, Shiota T, Qin J, Tsujino H, Stewart WJ, Thomas JD, Porqueddu M, White JA, Blackstone EH. Cosgrove-Edwards Annuloplasty System: midterm results. Ann Thorac Surg. 2000 Mar;69(3):717-21. doi: 10.1016/s0003-4975(99)01543-x. PMID 10750749
- [Background] Chee T, Haston R, Togo A, Raja SG. Is a flexible mitral annuloplasty ring superior to a semi-rigid or rigid ring in terms of improvement in symptoms and survival? Interact Cardiovasc Thorac Surg. 2008 May;7(3):477-84. doi: 10.1510/icvts.2007.174243. Epub 2008 Mar 4. PMID 18319323
- [Background] Meyer MA, von Segesser LK, Hurni M, Stumpe F, Eisa K, Ruchat P. Long-term outcome after mitral valve repair: a risk factor analysis. Eur J Cardiothorac Surg. 2007 Aug;32(2):301-7. doi: 10.1016/j.ejcts.2007.05.008. Epub 2007 Jun 11. PMID 17561410
- [Background] Chang BC, Youn YN, Ha JW, Lim SH, Hong YS, Chung N. Long-term clinical results of mitral valvuloplasty using flexible and rigid rings: a prospective and randomized study. J Thorac Cardiovasc Surg. 2007 Apr;133(4):995-1003. doi: 10.1016/j.jtcvs.2006.10.023. Epub 2007 Feb 22. PMID 17382640
- [Background] Staniloae C, Dupuis J, White M, Gosselin G, Dyrda I, Bois M, Crepeau J, Bonan R, Caron A, Lavoie J. Reduced pulmonary clearance of endothelin in congestive heart failure: a marker of secondary pulmonary hypertension. J Card Fail. 2004 Oct;10(5):427-32. doi: 10.1016/j.cardfail.2004.01.008. PMID 15470654
- See also: Related Info — http://www.micardia.com